CLINICAL TRIAL: NCT02585570
Title: Effect of Phenylephrine Infusion for Preventing Hypotension During Shoulder Arthroscopic Surgery in the Beach Chair Position
Brief Title: Effect of Phenylephrine During Shoulder Arthroscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Ki Hwa Lee, Assistant professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015-096
Record Dates: First submitted 2015-10-19; First posted 2015-10-23 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Disorder of Shoulder; Anesthesia
Keywords: shoulder; phenylephrine; hypotension
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose phenylephrine (Experimental): phenylephrine 0.5 mcg/kg/min
  Interventions: Drug: Phenylephrine
- High dose phenylephrine (Experimental): phenylephrine 1.0 mcg/kg/min .
  Interventions: Drug: Phenylephrine
- Normal saline (No Intervention): normal saline for 5minutes

INTERVENTIONS:
Drug: Phenylephrine — Patients is received phenylephrine 1.0 mcg/kg/min or 0.5 mcg/kg/min for 5 minutes before being placed in the beach chair position.
  Other Names: Phenylephrine hydrochloride
  Arms: High dose phenylephrine; Low dose phenylephrine

SUMMARY:
The purpose of this study is to determine whether phenylephrine infusion are effective in the prevention of hypotension after changing position to beach chair position during general anesthesia for shoulder arthroscopic surgery.

Investigators hypothesized that by increasing arterial blood pressure with phenylephrine infusion, incidence of hypotension would be decreased.

DETAILED DESCRIPTION:
The beach chair position is associated with hypotension, risk of cerebral hypoperfusion, and cerebral injury. Sixty-six patients undergoing elective shoulder arthroscopic surgery are randomized to receive either phenylephrine low dose (0.5 mcg/kg/hr), phenylephrine high dose (1.0 mcg/kg/min), or normal saline 5 minute before being placed in the beach chair position.

General anesthesia is induced with propofol, remifentanil and rocuronium (0.6 mg/kg) and the trachea intubated. Anesthesia is maintained with sevoflurane and remifentanil targeting for a BIS value 40-60. After hemodynamic stabilization, patients received on infusion of either phenylephrine high dose (1.0 mcg/kg/min), phenylephrine low dose (0.5 mcg/kg/hr) or normal saline 5 minute before being placed in the beach chair position. Following 15 minutes of infusion study drugs, measurements of mean arterial blood pressure and cardiac function (stroke volume variation, stroke volume index, and cardiac index) using Vigileo/Flotrac system were made.

ELIGIBILITY:
Inclusion Criteria:

* shoulder arthroscopic surgery undergone beach chair position

Exclusion Criteria:

* History of cerebrovascular event,
* significant cardiac disease (New York Heart Association symptoms class ≥ 3)
* uncontrolled hypertensive patients.
* American society of anesthesiologist class 4,5

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | 30 minutes
  After being beach chair position during shoulder arthroscopic surgery. We measure the incidence of hypotension with invasive blood pressure (Arterial line catheterization).

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hwa Lee, M.D, Principal Investigator — Haeundae paik hospital, inje university
Locations (1):
- Haeundae paik hospital, inje university, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soeding PF, Hoy S, Hoy G, Evans M, Royse CF. Effect of phenylephrine on the haemodynamic state and cerebral oxygen saturation during anaesthesia in the upright position. Br J Anaesth. 2013 Aug;111(2):229-34. doi: 10.1093/bja/aet024. Epub 2013 Mar 21. PMID 23518801